## EFFECTIVENESS OF NEGATIVE-PRESSURE WOUND THERAPY COMPARED TO WET-DRY DRESSING IN PRESSURE INJURIES

**Date of document** 

03.03.2020

**ICF** 

**Informed Consent Form** 

Study Title: Effectiveness of negative-pressure wound therapy compared to wet-dry dressing

in pressure injuries

Investigator: Ezgi Şahin

Study Director 1. Selda Rızalar

Study Director 2. Emre Özker

Dear participant,

This study aimed to determine the effect of topical negative pressure therapy on healing and cost in pressure injuries. Topical Negative Pressure therapy is a therapeutic vacuum wound closure method used to advance wound healing III. or IV. Stage. You are asked to participate in this research because you have a stage pressure wound. After accepting to participate in the research in writing, you are expected to answer the questions in the data collection form to learn general information about you. Wound healing will be evaluated with the 3D Wound Area, Volume, Tissue Classification Device and Pressure Ulcer Healing Assessment Scale to follow the improvements in your pressure wound healing. Only the wound area will be photographed with the help of the device following the healing of your wound. The dimensions (size, borders and depth) of your pressure wound will be measured. You are free to take part in this research or not. Participation in the study is voluntary. You can refuse to participate in this study. Participating in this research is entirely voluntary, and if you refuse it, any there will be no change. You also have the right to withdraw your consent at any stage of the study. You will not be charged for this therapy and care. You will not receive an additional payment because you have participated in the study. These records we obtained can be used in education or scientific publications in the field of health without stating your identity. Apart from these purposes, these records will not be used and will not be given to others. Thanks in advance for

Ezgi Şahin

Tel: 0 216 554 15 00

e.mail: earayan84@gmail.com

your participation and support.

Patient's Declaration

I was invited by Nurse Ezgi ŞAHİN as a "participant" to the research "The Effect of Topical

Negative Pressure Therapy on Healing and Cost" in Pressure Ulcers. I have been given

sufficient confidence that my personal information will be protected during the use of research

results for educational and scientific purposes. During the research, I can withdraw from the

research at any time without giving any reason. I don't assume any monetary responsibility for

the expenditures for the research. I will not receive a payment.

During the research, when I encounter a problem related to the pressure applied treatment; I

know that I can call researcher Ezgi Şahin on 0216 554 15 00.

I don't have to participate in this research and may not participate. I did not encounter any

compulsive behavior in participating in the research. I know that if I refuse to participate, this

will not harm my medical care. I understand all the explanations made to me in detail.

I decided to take part in this research project mentioned as a "participant" after a certain period

of thinking on my own.

I voluntarily accept the work done on this subject.

Date:

Patient Name Surname:

Signature: